CLINICAL TRIAL: NCT05839691
Title: Improving the Cardiovascular Health of High-Risk Families Through an Innovative Home Visitation Intervention
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Gareth R. Dutton PhD, Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300008424; UG3HL162973 (NIH)
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Nutrition, Healthy; Maternal Behavior; Health Behavior
Keywords: Home Visiting Program
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mothers: Mothers enrolled in Home Visiting Programs that have or will be participating in past or future projects.
- Home Visitors: Home Visitors/Educators employed by Home Visiting Programs that have or will be participating in past or future projects.
- Supervisors: Supervising staff of Home Visiting Programs that have or will be participating in past or future projects.

SUMMARY:
The purpose of this study is to conduct formative work with relevant stakeholders, including families and home visitation program staff involved in previous studies and/or future projects, to understand facilitators, barriers, and other attitudes related to incorporating cardiovascular health topics into existing curricula and to obtain input on treatment modifications for future programs.

DETAILED DESCRIPTION:
Alabama Department of Early Childhood Education administers an annual electronic survey to all home-visiting program staff and enrolled families. The survey queries these individuals about demographics, program satisfaction, and interest in new programming. We will request deidentified survey data to understand what proportion of families currently being served are currently expecting (pregnant) or are within one year post-partum. Those that fall in that category will be asked survey questions gauging their interest in cardiovascular health topics. Additionally, home-visiting staff will be asked about their comfort-level discussing the cardiovascular health topics with their clients. Home-visiting program staff will also be invited to participate in group-setting qualitative interviews focused on facilitators, barriers, and other attitudes related to any new programming or material related to cardiovascular health topics in the future. Interviews will be audio-recorded, transcribed verbatim, and the file will be erased after the transcripts have been verified for completeness. The transcription will not have any identifiable data included as participants will use anonymous names or nicknames and/or their study identification number during the interview sessions.

ELIGIBILITY:
Inclusion Criteria:

- capable and willing to complete an electronic survey and/or an online group interview via Zoom

AND

* participants must be an expectant mother (currently pregnant) OR
* a mother within one year of giving birth AND
* currently enrolled in a partner home-visiting program

OR

- participants are an employee of a partner home-visiting program

Exclusion Criteria:

- individuals are not an employee of a partner home-visiting program

Nor

* an expectant mother (currently pregnant) or within one year of giving birth AND
* not currently enrolled in a partner home-visiting program

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mothers currently pregnant or within one year of giving birth currently enrolled in a partner home-visiting program and employees of partner home-visiting programs
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Home Visiting Caregivers who are pregnant or within one-year post delivery | At Enrollment
  Percentage of survey respondents (out of total respondents) who self-report they are currently pregnant or gave birth within the last year. Participants will self-report by responding to a one-item, multiple choice survey question. In response, they can mark all that apply of the following: a) I am currently pregnant, b) I gave birth to a child who currently is less than 6 months old, c) I gave birth to a child who is currently between 6 months and less than 1 year old, d) I gave birth to a child who is currently between 1 year and 2 years old, e) None of these apply to me

SECONDARY OUTCOMES:
Comfort level of home visiting staff discussing eating healthy with home visiting clients. | At Enrollment
  Proportion of respondents responding very uncomfortable vs uncomfortable vs neither comfortable nor uncomfortable vs comfortable vs very comfortable with "very comfortable" indicating the most comfort to the following question: how comfortable are you discussing eating healthy with your home visiting clients?
Comfort level of home visiting staff discussing being more active with home visiting clients. | At Enrollment
  Proportion of respondents responding very uncomfortable vs uncomfortable vs neither comfortable nor uncomfortable vs comfortable vs very comfortable with "very comfortable" indicating the most comfort with "very comfortable" indicating the most comfort to the following question: how comfortable are you discussing being more active with your home visiting clients?
Comfort level of home visiting staff discussing getting healthy sleep with home visiting clients. | At Enrollment
  Proportion of respondents responding very uncomfortable vs uncomfortable vs neither comfortable nor uncomfortable vs comfortable vs very comfortable with "very comfortable" indicating the most comfort to the following question: how comfortable are you discussing getting healthy sleep with your home visiting clients?
Comfort level of home visiting staff discussing weight management with home visiting clients. | At Enrollment
  Proportion of respondents responding very uncomfortable vs uncomfortable vs neither comfortable nor uncomfortable vs comfortable vs very comfortable with "very comfortable" indicating the most comfort to the following question: how comfortable are you discussing weight management with your home visiting clients?
Comfort level of home visiting staff discussing stress management with home visiting clients. | At Enrollment
  Proportion of respondents responding very uncomfortable vs uncomfortable vs neither comfortable nor uncomfortable vs comfortable vs very comfortable with "very comfortable" indicating the most comfort to the following question: how comfortable are you discussing stress management with your home visiting clients?
Comfort level of home visiting staff discussing quitting tobacco with home visiting clients. | At Enrollment
  Proportion of respondents responding very uncomfortable vs uncomfortable vs neither comfortable nor uncomfortable vs comfortable vs very comfortable with "very comfortable" indicating the most comfort to the following question: how comfortable are you discussing quitting tobacco with your home visiting clients?
Comfort level of home visiting staff discussing controlling cholesterol with home visiting clients. | At Enrollment
  Proportion of respondents responding very uncomfortable vs uncomfortable vs neither comfortable nor uncomfortable vs comfortable vs very comfortable with "very comfortable" indicating the most comfort to the following question: how comfortable are you discussing controlling cholesterol with your home visiting clients?
Comfort level of home visiting staff discussing managing blood sugar with home visiting clients. | At Enrollment
  Proportion of respondents responding very uncomfortable vs uncomfortable vs neither comfortable nor uncomfortable vs comfortable vs very comfortable with "very comfortable" indicating the most comfort to the following question: how comfortable are you discussing managing blood sugar with your home visiting clients?
Comfort level of home visiting staff discussing managing blood pressure with home visiting clients. | At Enrollment
  Proportion of respondents responding very uncomfortable vs uncomfortable vs neither comfortable nor uncomfortable vs comfortable vs very comfortable with "very comfortable" indicating the most comfort to the following question: how comfortable are you discussing managing blood pressure with your home visiting clients?

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Dutton, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States